CLINICAL TRIAL: NCT06597682
Title: A Randomized Controlled Basket Study for Evaluating Immunomodulatory Interventions in Post-Acute Sequelae of SARS-CoV-2 InfEction (RISE)
Brief Title: Evaluating Immunomodulatory Interventions in Post-Acute Sequelae of SARS-CoV-2 InfEction
Acronym: RISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RISE
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-01

CONDITIONS: Post-acute Sequelae of SARS-COV-2 Infection
Keywords: Post-acute Sequelae of SARS-COV-2 Infection; Long COVID; Immunomodulatory Interventions
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Prednisone; Budesonide, Formoterol Fumarate Drug Combination; montelukast; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Inflammatory Cardiac Involvement symptom cluster - immunomodulatory intervention (Experimental)
  Interventions: Drug: Prednisone; Drug: Vitamin C combined with Coenzyme Q10 oral treatment
- Inflammatory Cardiac Involvement symptom cluster (Active Comparator)
  Interventions: Drug: Vitamin C combined with Coenzyme Q10 oral treatment
- Cough symptom cluster - immunomodulatory intervention (Experimental)
  Interventions: Drug: Budesonide/Formoterol; Drug: Montelukast tablets oral treatment
- Cough symptom cluster (Active Comparator)
  Interventions: Drug: Montelukast tablets oral treatment
- Fatigue symptom cluster - immunomodulatory intervention (Experimental)
  Interventions: Drug: Prednisone; Drug: Vitamin C combined with Coenzyme Q10 oral treatment
- Fatigue symptom cluster (Active Comparator)
  Interventions: Drug: Vitamin C combined with Coenzyme Q10 oral treatment

INTERVENTIONS:
Drug: Prednisone — Total 4 weeks of treatment
  Arms: Fatigue symptom cluster - immunomodulatory intervention; Inflammatory Cardiac Involvement symptom cluster - immunomodulatory intervention
Drug: Budesonide/Formoterol — Total 8 weeks of treatment
  Arms: Cough symptom cluster - immunomodulatory intervention
Drug: Vitamin C combined with Coenzyme Q10 oral treatment — Total 4 weeks of treatment
  Arms: Fatigue symptom cluster; Fatigue symptom cluster - immunomodulatory intervention; Inflammatory Cardiac Involvement symptom cluster; Inflammatory Cardiac Involvement symptom cluster - immunomodulatory intervention
Drug: Montelukast tablets oral treatment — Total 8 weeks of treatment
  Arms: Cough symptom cluster; Cough symptom cluster - immunomodulatory intervention

SUMMARY:
This study is a prospective, randomized controlled, basket trial. Patients diagnosed with Post-Acute Sequelae of SARS-CoV-2 Infection who meet the inclusion and exclusion criteria are recruited and divided into three symptom clusters: Inflammatory Cardiac involvement symptoms cluster, cough symptoms cluster and fatigue symptoms cluster. Each symptom cluster is randomly divided into an experimental group and a control group, Patients who do not accept treatment can be included in the observational cohort. Subjects in the experimental group receive immunomodulatory interventions plus conventional treatment, while subjects in the control group receive conventional treatment only. Subjects in each symptom cluster undergo clinical medical record data collection, laboratory tests, and imaging examinations at specified time points, as well as records of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years;
* 2. Post-infection with SARS-CoV-2 for more than 3 months and meets the World Health Organization (WHO) definition of Long COVID;
* 3. Symptom criteria: Meet the inclusion and exclusion criteria for each symptom cluster;
* 4. Fertile female subjects are not breastfeeding or pregnant at the time of enrollment (negative urine pregnancy test);
* 5. Willing and able to provide informed consent, complete surveys, clinical assessments, and all necessary follow-up visits;

Symptom Cluster Inclusion Criteria:

* Inflammatory Cardiac Involvement Symptom Cluster
* 1) Age: 18-75 years old;
* 2) Presence of cardiac symptoms at the time of enrollment (e.g., Chest tightness after physical activity, chest pain, difficulty breathing, palpitations, fatigue, etc.);
* 3) CMR shows the following abnormal findings based on any of the following criteria:
* a) Native T1 increase ≥ 1130 milliseconds at 3.0 T (or an increase of 1030 milliseconds at 1.5 T) and/or;
* b) Native T2 ≥ 39.5 milliseconds at 3.0 T (or 49.5 milliseconds at 1.5 T) and/or;
* c) Presence of non-ischemic myocardial and pericardial late gadolinium enhancement and/or;
* d) Left ventricular ejection fraction ≥ 40% and ≤50%.
* Cough Symptom Cluster
* 1) Clinical assessment of cough according to ACCP guidelines indicates no cough caused by other diseases such as COPD, asthma, chronic bronchitis, gastroesophageal reflux, bronchiectasis, etc.;
* 2) Chest X-ray or CT scan shows no abnormalities that could lead to cough or other serious lung diseases;
* 3) FENO ≥25 ppb, or the proportion of eosinophils in sputum cytology ≥2.5%; or the blood eosinophil count >0.3×10⁹/L.
* Fatigue Symptom Cluster
* 1) Fatigue Severity Scale (FSS) average score ≥ 4;
* 2) Any inflammatory marker (CRP, ESR, PCT, ferritin, IL-6, TNFα) is above the upper limit of normal.

Exclusion Criteria:

* 1. Known SARS-CoV-2 infection within 3 months prior to the date of informed consent signature;
* 2. Systemic fungal infection and active infections that cannot be controlled by anti-infective agents;
* 3. Current or recent (within the last 10 weeks) use of glucocorticoids, other immunosuppressants, or biologic agents;
* 4. Known allergy/sensitivity or any hypersensitivity reaction to the study intervention or control components;
* 5. Known contraindications to the study intervention;
* 6. Any persistent central nervous system disorders, psychiatric illnesses, chronic respiratory or cardiac diseases, Underlying diseases (poorly controlled diabetes, poorly controlled hypertension, peripheral edema, cataracts or glaucoma, peptic ulcer disease, femoral head necrosis, low bone density, or osteoporosis);
* 7. For female participants: pregnant or breastfeeding at screening, or expecting to become pregnant during the study period; women of childbearing age who are unwilling to use effective contraceptive measures (defined as PEARL index <1, such as birth control pills, intrauterine devices);
* 8. Known alcohol, drug, or chemical abuse;
* 9. Currently participating in another clinical trial;
* 10. Deemed ineligible to participate in this study by the investigator's assessment.

Symptom Cluster Exclusion Criteria:

* Inflammatory Cardiac Involvement Symptom Cluster
* 1) Past medical history or cardiac magnetic resonance (CMR) evidence indicating significant cardiac disease, including:
* a) Known left ventricular ejection fraction (LVEF) <40% indicating cardiac dysfunction;
* b) Congestive heart failure (New York Heart Association Class III-IV);
* c) Ongoing treatment for heart failure (including HFrEF and HFpEF);
* d) Confirmed ischemic heart disease, peripheral artery disease, and/or cerebrovascular disease;
* e) Persistent or permanent atrial fibrillation or significant arrhythmias;
* f) Congenital or clinically relevant valvular heart disease (moderate or severe);
* g) Specific cardio myopathies (hypertrophic, hypertensive heart disease, amyloidosis, previous myocarditis, non-ischemic dilated cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, non-compacted cardiomyopathy, etc.);
* 2) Contraindications for contrast-enhanced cardiac magnetic resonance (CMR) imaging, such as: use of implanted devices not compatible with MRI; known allergy to gadolinium-based contrast agents (CBGA);
* 3) Patients with structural heart disease or incidental arrhythmias detected on cardiac magnetic resonance imaging will be advised to consult their physicians.
* Cough Symptom Cluster
* 1) Current smoker or having quit smoking for less than 6 months;
* 2) Intolerance to pulmonary function testing and/or FeNO;
* 3) Chest CT showing acute pulmonary infection-related diseases;
* 4) Forced expiratory volume in 1 second (FEV1) / Forced vital capacity (FVC) ratio less than 60%;
* 5) Currently taking or having used angiotensin-converting enzyme inhibitors (ACEI) within the past 3 months of screening;
* 6) Received any relevant traditional Chinese or Western medical treatment within the last month.
* Fatigue Symptom Cluster
* 1) Received any relevant traditional Chinese or Western medical treatment within the last month, taking sedatives, hypnotics, melatonin, or antidepressants;
* 2) Known previous diagnosis of myalgic encephalomyelitis/chronic fatigue syndrome unrelated to SARS-CoV-2 infection;
* 3) Known previous autonomic dysfunction unrelated to SARS-CoV-2 infection;
* 4) Fatigue caused by metabolism-related diseases (such as hyperthyroidism or hypothyroidism, malnutrition) that developed following SARS-CoV-2 infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Cardiac Involvement symptom cluster: cardiac magnetic resonance (CMR) indicators | 4 weeks
  Assessing the difference in changes in cardiac magnetic resonance (CMR) indicators [left ventricular ejection fraction, late gadolinium enhancement (LGE), and T1 and T2 mapping values (in milliseconds)] from baseline between the experimental and control groups.
Cough symptom cluster: Leicester Cough Questionnaire (LCQ) scale scores | 8 weeks
  Assessing the difference in changes in the Leicester Cough Questionnaire (LCQ) scale scores from baseline.
  The total score range of the LCQ is from 3 to 21 points, with higher scores indicating a lesser impact of cough on the patient's life.
Fatigue symptom cluster: Fatigue Severity Scale (FSS) scale scores | 4 weeks
  Assessing the difference in changes in the Fatigue Severity Scale (FSS) scale scores from baseline.
  The total score range of the FSS is from 9 to 63 points, with higher scores indicating a greater severity of fatigue.

SECONDARY OUTCOMES:
Inflammatory Cardiac Involvement symptom cluster: other relevant cardiac magnetic resonance (CMR) indicators | 4 weeks
  Assessing the changes in in other relevant cardiac magnetic resonance (CMR) indicators from baseline.
Inflammatory Cardiac Involvement symptom cluster: VO2max | At baseline, 4 weeks
  Assessing the changes in VO2max in cardiopulmonary exercise testing.
Inflammatory Cardiac Involvement symptom cluster: Kansas City Cardiomyopathy Questionnaire (KCCQ) scores | At baseline, 4, 8, 12, and 24 weeks
  Assessing the changes in the KCCQ scores between the experimental and control groups.
  The total score range of the KCCQ is from 0 to 100, with lower scores indicating poorer quality of life for heart failure patients.
Inflammatory Cardiac Involvement symptom cluster: Change in cTNT Levels | At baseline, 4, 8, 12 and 24 weeks
  Measures the change in cardiac troponin T (cTNT) levels
Inflammatory Cardiac Involvement symptom cluster: the proportion of patients experiencing heart failure and major adverse cardiac events (MACE) | From baseline to 52 weeks
  From baseline to week 52, assessing the proportion of patients experiencing heart failure and MACE between the experimental and control groups.
EuroQoL 5-Dimension 5-Level (EQ-5D-5L) questionnaire scores | At baseline, 4, 8, 12 and 24 weeks
  Assessing the changes in the EQ-5D-5L questionnaire scores between the experimental and control groups.
  The EQ-5D-5L is a widely used generic measure of health status consisting of two parts.
  The first part (the descriptive system) provides a descriptive profile that can be used to generate a health state profile. Each health state can be assigned a summary index score. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
  The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Pittsburgh Sleep Quality Index (PSQI) scores | At baseline 4, 8, 12, and 24 weeks
  Assessing the changes in the PSQI scores between the experimental and control groups.
  The total score range of the PSQI is from 0 to 21, with higher scores indicating poorer sleep quality.
Generalized Anxiety Disorder-7 (GAD-7) | At baseline, 4, 8, 12 and 24 weeks
  Assessing the changes in the GAD-7 scores between the experimental and control groups.
  The total score range of the GAD-7 is from 0 to 21, with higher scores indicating more severe anxiety.
Patient Health Questionnaire-9 (PHQ-9) depression symptom cluster scores | At baseline, 4, 8, 12 and 24 weeks
  Assessing the changes in the PHQ-9 cores between the experimental and control groups.
  The total score range of the PHQ-9 is from 0 to 27, with higher scores indicating more severe depression.
Cough symptom cluster: Visual Analogue Scale (VAS) | At baseline 4, 8 and 12 weeks
  Assessing the change in the severity of cough as measured by the VAS between the experimental and control groups .
  The total score range of the VAS is from 0 to 100, with higher scores indicating more severe coughing in the patient.
Cough symptom cluster: pulmonary function and fractional exhaled nitric oxide (FeNO) levels | At baseline and 8 weeks
  Assessing the changes in pulmonary function and FeNO levels between the experimental and control groups.
Fatigue symptom cluster: Visual Analogue Scale (VAS) | At baseline, 4, 8, and 12 weeks
  The total score range of the VAS is from 0 to 100, with higher scores indicating more severe fatigue in the patient.
Change in proBNP Levels | Baseline, 4, 8, 12, 24 weeks
  Measures the change in N-terminal pro-brain natriuretic peptide (proBNP) levels, which are associated with heart failure.
Change in Angiotensin II Levels | Baseline, 4, 8, 12, 24 weeks
  Measures the change in angiotensin II levels
Change in Ferritin Levels | Baseline, 4, 8, 12, 24 weeks
  Measures the change in ferritin levels
Change in IL-6 Levels | Baseline, 4, 8, 12, 24 weeks
  Measures the change in interleukin-6 (IL-6) levels
Change in hsCRP Levels | Baseline, 4, 8, 12, 24 weeks
  Measures the change in high-sensitivity C-reactive protein (hsCRP) levels

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No